CLINICAL TRIAL: NCT00000129
Title: Prospective Evaluation of Radial Keratotomy (PERK) Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: NEI-28
Record Dates: First submitted 1999-09-23; First posted 1999-09-24 (Estimated); Last update posted 2009-09-17 (Estimated); Status verified 2009-09

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Keratotomy, Radial

INTERVENTIONS:
Procedure: Radial Keratotomy

SUMMARY:
To determine whether radial keratotomy is effective in reducing myopia.

To detect complications of the surgery.

To discover patient characteristics and surgical factors affecting the results.

To determine the long-term safety and efficacy of the procedure.

DETAILED DESCRIPTION:
Approximately 11 million Americans have myopia that can be corrected with eyeglasses or contact lenses. Some of these people may also be candidates for radial keratotomy (RK), a procedure that aims to correct or reduce myopia by surgery that flattens the corneal curvature.

Keratotomy was first performed by surgeons in Europe and the United States in the late 1800s, and the basic optical and mechanical principles of the operation were defined in the 1940s and 1950s by the Japanese doctors T. Sato and K. Akiyama, who used anterior and posterior corneal incisions. The posterior incisions damaged the cornea, and the procedure was modified in the Soviet Union by doctors Fyodorov and V. Durnev to include incisions in only the anterior cornea. Since its introduction into the United States in 1978, numerous ophthalmologists have modified the procedure by introducing technical and surgical improvements such as ultrasonic methods to measure the thickness of the cornea and the use of diamond-bladed micrometer knives to make the incisions.

However, scientific assessment of RK lagged behind growing public and professional interest in the procedure. In 1980, in response to widespread concern about the long-term safety and efficacy of RK, a group of ophthalmic surgeons approached the National Eye Institute with a proposal for a multicenter clinical trial that would evaluate the potential benefits and risks of this procedure.

The Prospective Evaluation of Radial Keratotomy study, involving 435 patients and 99 pilot patients, was a clinical trial designed to evaluate the short- and long-term safety and efficacy of one technique of radial keratotomy. The procedure was evaluated by comparing a patient's refractive error and uncorrected vision before and after surgery. The more myopic eye received surgery first. Patients were required to wait 1 year before having the operation on the second eye.

The surgical technique was standardized, consisting of eight centrifugal radial incisions made manually with a diamond micrometer knife. The diameter of the central, uncut, clear zone was determined by the preoperative spherical equivalent cycloplegic refraction (-2.00 to -3.12 D = 4.0 mm; -3.25 to -4.3 D = 3.5 mm; -4.50 to -8.00 D = 3.0 mm). The blade length, which determined the depth of the incision, was set at 100 percent of the thinnest of four intraoperative ultrasonic corneal thickness readings taken paracentrally at the 3-, 6-, 9-, and 12-o'clock meridians just outside the mark delineating the clear zone. The incisions were made from the edge of the trephine mark to the limbal vascular arcade and were spaced equidistantly around the cornea.

Patients were examined preoperatively and after surgery at 2 weeks, 3 months, 6 months, annually for 5 years, and at 10 years. Examinations in the morning and evening of the same day were done at 3 months, 1 year, 3 years, and 11 years in a subset of the patients to test for diurnal fluctuation of vision and refraction.

The primary outcome variables measured at each visit was the uncorrected and spectacle-corrected visual acuity and the refractive error with the pupil dilated and undilated. The corneal shape was measured with central keratometry and photokeratoscopy. Endothelial function was evaluated using specular microscopy. A slit-lamp microscope examination was made to check for complications from the incisions. Contrast sensitivity was tested in a subset of patients. Patient motivation and satisfaction were studied with psychometric questionnaires at baseline, 1 year, 5-6 years, and 10 years.

ELIGIBILITY:
All men and women had 2 to 8 diopters of simple myopia and were correctable to 20/20 or better with glasses or contact lenses. All patients had the stability of their myopia documented by previous records. Patients were at least 21 years of age and lived in the metropolitan area of the study centers. Each patient agreed to have surgery on one eye and to wait 1 year for surgery on the other eye. Patients with systemic diseases that might affect corneal wound healing and patients with high corneal astigmatism were excluded from the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1981-04; Study Completion 1983-10 (Actual)

REFERENCES:
- [Background] Waring GO 3rd, Moffitt SD, Gelender H, Laibson PR, Lindstrom RL, Myers WD, Obstbaum SA, Rowsey JJ, Safir A, Schanzlin DJ, Bourque LB. Rationale for and design of the National Eye Institute Prospective Evaluation of Radial Keratotomy (PERK) Study. Ophthalmology. 1983 Jan;90(1):40-58. doi: 10.1016/s0161-6420(83)34603-0. PMID 6338438
- [Background] Bourque LB, Rubenstein R, Cosand B, Waring GO 3rd, Moffitt S, Gelender H, Laibson PR, Lindstrom RL, McDonald M, Myers WD, et al. Psychosocial characteristics of candidates for the prospective evaluation of radial keratotomy (PERK) study. Arch Ophthalmol. 1984 Aug;102(8):1187-92. doi: 10.1001/archopht.1984.01040030965027. PMID 6380467
- [Background] Novak AF; Lindstrom RL; Williams PA; Everson M; Corneal pachymetry prior to radial keratotomy: a comparison of techniques., J Refract Surg 1985;1:151-153
- [Background] Steinberg EB, Waring GO 3rd. Comparison of two methods of marking the visual axis on the cornea during radial keratotomy. Am J Ophthalmol. 1983 Nov;96(5):605-8. doi: 10.1016/s0002-9394(14)73417-8. PMID 6638126
- [Background] Steinberg EB, Wilson LA, Waring GO 3rd, Lynn MJ, Coles WH. Stellate iron lines in the corneal epithelium after radial keratotomy. Am J Ophthalmol. 1984 Oct 15;98(4):416-21. doi: 10.1016/0002-9394(84)90122-3. PMID 6486212
- [Background] Nelson JD, Williams P, Lindstrom RL, Doughman DJ. Map-fingerprint-dot changes in the corneal epithelial basement membrane following radial keratotomy. Ophthalmology. 1985 Feb;92(2):199-205. doi: 10.1016/s0161-6420(85)34055-1. PMID 3872431
- [Background] Waring GO 3rd, Lynn MJ, Gelender H, Laibson PR, Lindstrom RL, Myers WD, Obstbaum SA, Rowsey JJ, McDonald MB, Schanzlin DJ, et al. Results of the prospective evaluation of radial keratotomy (PERK) study one year after surgery. Ophthalmology. 1985 Feb;92(2):177-98, 307. doi: 10.1016/s0161-6420(85)34054-x. PMID 3885128
- [Background] Atkin A, Asbell P, Justin N, Smith H, Wayne R, Winterkorn J. Radial keratotomy and glare effects on contrast sensitivity. Doc Ophthalmol. 1986 Feb 28;62(2):129-48. doi: 10.1007/BF00229125. PMID 3956364
- [Background] Bourque LB, Cosand BB, Drews C, Waring GO 3rd, Lynn M, Cartwright C. Reported satisfaction, fluctuation of vision, and glare among patients one year after surgery in the Prospective Evaluation of Radial Keratotomy (PERK) Study. Arch Ophthalmol. 1986 Mar;104(3):356-63. doi: 10.1001/archopht.1986.01050150056026. PMID 3954634
- [Background] Bourque LB; Cosand BB; Drews C; Waring GO; Lynn M; Cartwright C; Satisfaccion informada, fluctuacion de la vision y resplandor en pacientes al cabo de un ano tras la cirugia en el estudio de la evaluacion prospectiva de la queratotomia radial (EPQR)., Arch Ophthalmol 1986;2:57-64
- [Background] Mandelbaum S, Waring GO 3rd, Forster RK, Culbertson WW, Rowsey JJ, Espinal ME. Late development of ulcerative keratitis in radial keratotomy scars. Arch Ophthalmol. 1986 Aug;104(8):1156-60. doi: 10.1001/archopht.1986.01050200062050. PMID 3741245
- [Background] Schanzlin DJ, Santos VR, Waring GO 3rd, Lynn M, Bourque L, Cantillo N, Edwards MA, Justin N, Reinig J, Roszka-Duggan V. Diurnal change in refraction, corneal curvature, visual acuity, and intraocular pressure after radial keratotomy in the PERK Study. Ophthalmology. 1986 Feb;93(2):167-75. doi: 10.1016/s0161-6420(86)33765-5. PMID 3951823
- [Background] Villasenor RA, Santos VR, Cox KC, Harris DF 2nd, Lynn M, Waring GO 3rd. Comparison of ultrasonic corneal thickness measurements before and during surgery in the prospective evaluation of Radial Keratotomy (PERK) Study. Ophthalmology. 1986 Mar;93(3):327-30. doi: 10.1016/s0161-6420(86)33746-1. PMID 3517739
- [Background] Lynn MJ; Waring GO; Predictability and stability of radial keratotomy., J. Refract Surg 1987;3:193-196
- [Background] Lynn MJ, Waring GO 3rd, Sperduto RD. Factors affecting outcome and predictability of radial keratotomy in the PERK Study. Arch Ophthalmol. 1987 Jan;105(1):42-51. doi: 10.1001/archopht.1987.01060010048030. PMID 3800746
- [Background] Santos VR, Waring GO 3rd, Lynn MJ, Holladay JT, Sperduto RD. Relationship between refractive error and visual acuity in the Prospective Evaluation of Radial Keratotomy (PERK) Study. Arch Ophthalmol. 1987 Jan;105(1):86-92. doi: 10.1001/archopht.1987.01060010092038. PMID 3800751
- [Background] Waring GO 3rd, Lynn MJ, Culbertson W, Laibson PR, Lindstrom RD, McDonald MB, Myers WD, Obstbaum SA, Rowsey JJ, Schanzlin DJ. Three-year results of the Prospective Evaluation of Radial Keratotomy (PERK) Study. Ophthalmology. 1987 Oct;94(10):1339-54. doi: 10.1016/s0161-6420(87)80021-0. PMID 3684210
- [Background] Cartwright CS, Bourque LB, Lynn M, Waring GO 3rd. Relationship of glare to uncorrected visual acuity and cycloplegic refraction 1 year after radial keratotomy in the prospective evaluation of radial keratotomy (PERK) study. J Am Optom Assoc. 1988 Jan;59(1):36-9. PMID 3278044
- [Background] McDonnell PJ, Schanzlin DJ. Early changes in refractive error following radial keratotomy. Arch Ophthalmol. 1988 Feb;106(2):212-4. doi: 10.1001/archopht.1988.01060130222031. PMID 3341977
- [Background] Rowsey JJ, Balyeat HD, Monlux R, Holladay J, Waring GO 3rd, Lynn MJ. Prospective evaluation of radial keratotomy. Photokeratoscope corneal topography. Ophthalmology. 1988 Mar;95(3):322-34. doi: 10.1016/s0161-6420(88)33179-9. PMID 3174000
- [Background] Santos VR, Waring GO 3rd, Lynn MJ, Schanzlin DJ, Cantillo N, Espinal ME, Garbus J, Justin N, Roszka-Duggan V. Morning-to-evening change in refraction, corneal curvature, and visual acuity 2 to 4 years after radial keratotomy in the PERK Study. Ophthalmology. 1988 Nov;95(11):1487-93. doi: 10.1016/s0161-6420(88)32981-7. PMID 3211457
- [Background] Serle JB, Asbell PA, Obstbaum SA, Podos SM, Anh-Le N. The evaluation of corneal endothelial permeability in PERK study patients. Br J Ophthalmol. 1988 Apr;72(4):274-7. doi: 10.1136/bjo.72.4.274. PMID 3378023
- [Background] Lynn MJ, Waring GO 3rd, Nizam A, Kutner MH, Culbertson W, McDonald MB, Meyers WD, Naidoff MA, Nelson JD, Obstbaum SA, et al. Symmetry of refractive and visual acuity outcome in the Prospective Evaluation of Radial Keratotomy (PERK) study. Refract Corneal Surg. 1989 Mar-Apr;5(2):75-81. PMID 2488790
- [Background] Rowsey JJ, Monlux R, Balyeat HD, Stevens SX, Gelender H, Holladay J, Krachmer JH, Laibson P, Lindstrom R, Lynn M, et al. Accuracy and reproducibility of KeraScanner analysis in PERK corneal topography. PERK Study Group. Curr Eye Res. 1989 Jul;8(7):661-74. doi: 10.3109/02713688909025800. PMID 2791617
- [Background] Ginsburg AP, Waring GO 3rd, Steinberg EB, Williams PA, Justin N, Deitz JR, Roszka-Duggan VK, Baluvelt K, Bourque L. Contrast sensitivity under photopic conditions in the Prospective Evaluation of Radial Keratotomy (PERK) Study. Refract Corneal Surg. 1990 Mar-Apr;6(2):82-91. PMID 2248920
- [Background] Lynn MJ, Waring GO 3rd, Carter JT. Combining refractive error and uncorrected visual acuity to assess the effectiveness of refractive corneal surgery. Refract Corneal Surg. 1990 Mar-Apr;6(2):103-9; discussion 109-12. PMID 2248912
- [Background] Waring GO 3rd, Lynn MJ, Fielding B, Asbell PA, Balyeat HD, Cohen EA, Culbertson W, Doughman DJ, Fecko P, McDonald MB, et al. Results of the Prospective Evaluation of Radial Keratotomy (PERK) Study 4 years after surgery for myopia. Perk Study Group. JAMA. 1990 Feb 23;263(8):1083-91. PMID 2405203
- [Background] Holladay JT, Lynn MJ, Waring GO 3rd, Gemmill M, Keehn GC, Fielding B. The relationship of visual acuity, refractive error, and pupil size after radial keratotomy. Arch Ophthalmol. 1991 Jan;109(1):70-6. doi: 10.1001/archopht.1991.01080010072036. PMID 1987953
- [Background] Rowsey JJ, Waring GO 3rd, Monlux RD, Balyeat HD, Stevens SX, Culbertson W, Barron B, Nelson D, Asbell P, Smith R, et al. Corneal topography as a predictor of refractive change in the prospective evaluation of radial keratotomy (PERK) study. Ophthalmic Surg. 1991 Jul;22(7):370-80. PMID 1891181
- [Background] Waring GO 3rd, Lynn MJ, Nizam A, Kutner MH, Cowden JW, Culbertson W, Laibson PR, McDonald MB, Nelson JD, Obstbaum SA, et al. Results of the Prospective Evaluation of Radial Keratotomy (PERK) Study five years after surgery. The Perk Study Group. Ophthalmology. 1991 Aug;98(8):1164-76. doi: 10.1016/s0161-6420(91)32156-0. PMID 1923352
- [Background] Waring GO 3rd, Lynn MJ, Strahlman ER, Kutner MH, Culbertson W, Laibson PR, Linstrom RD, McDonald MB, Myers WD, Obstbaum SA, et al. Stability of refraction during four years after radial keratotomy in the prospective evaluation of radial keratotomy study. Am J Ophthalmol. 1991 Feb 15;111(2):133-44. doi: 10.1016/s0002-9394(14)72250-0. PMID 1801760
- [Background] Nizam A, Waring GO 3rd, Lynn MJ, Ward MA, Asbell PA, Balyeat HD, Cohen E, Culbertson W, Doughman DJ, Fecko P, et al. Stability of refraction and visual acuity during 5 years in eyes with simple myopia. The PERK Study Group. Refract Corneal Surg. 1992 Nov-Dec;8(6):439-47. PMID 1493117
- [Background] Bourque LB, Lynn MJ, Waring GO 3rd, Cartwright C. Spectacle and contact lens wearing six years after radial keratotomy in the Prospective Evaluation of Radial Keratotomy Study. Ophthalmology. 1994 Mar;101(3):421-31. doi: 10.1016/s0161-6420(94)31315-7. PMID 8127562
- [Background] Waring GO 3rd, Lynn MJ, McDonnell PJ. Results of the prospective evaluation of radial keratotomy (PERK) study 10 years after surgery. Arch Ophthalmol. 1994 Oct;112(10):1298-308. doi: 10.1001/archopht.1994.01090220048022. PMID 7945032
- [Background] McDonnell PJ, Nizam A, Lynn MJ, Waring GO 3rd. Morning-to-evening change in refraction, corneal curvature, and visual acuity 11 years after radial keratotomy in the prospective evaluation of radial keratotomy study. The PERK Study Group. Ophthalmology. 1996 Feb;103(2):233-9. doi: 10.1016/s0161-6420(96)30711-2. PMID 8594507
- [Background] Waring GO; Lynn MJ; McDonnell PJ; Resultados del estudio de evaluacion Prospectiva de la Queratotomia Radial (EPQR) 10 anos despues de la cirugia., Arch Ophthalmol (Edicion Espanola) 1995;6:99-110
- [Background] Nizam A; Waring GO; Lynn MJ; Stability of refraction during 11 years in eyes with simple myopia., Invest Ophthalmol Vis Sci 1996;37:S1004